CLINICAL TRIAL: NCT06574243
Title: Positive Education Through Social Media to Reduce Negative Stereotypes Towards Old Age: a Quasi-experimental Study
Brief Title: Positive Education Through Social Media to Reduce Negative Stereotypes Towards Old Age
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Elena de la Fuente, Doctor, Universidad de Zaragoza
Other Study IDs: U1111-1311-9233
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Ageism
Keywords: healthy aging; ageism; negative stereotypes; social media.
MeSH Terms: conditions — Ageism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Social media education — The intervention consisted of daily positive messages about aging posted on an Instagram account (@laetapaplateada), created specifically for this study, and was conducted over the course of a week. Examples included "The ability to make decisions improves with age" and "Emotional regulation improves with age" (David, 2017). These posts were accompanied by their respective author references

SUMMARY:
Introduction and Objectives: To assess the effectiveness of positive psychoeducation regarding aging, disseminated through social media channels, in mitigating negative stereotypes. Additionally, we aim to explore any potential associations between various sociodemographic variables and the prevalence of negative stereotypes towards the elderly.

Methods: This quasi-experimental study involved an experimental group comprising subjects who underwent a 7-day intervention. The study aimed to evaluate any alterations in negative stereotypes towards aging both before and after the intervention. The intervention consisted of daily publication of positive messages about aging on a social media account. Two questionnaires were used: one collecting sociodemographic variables and the Questionnaire for Evaluating Negative Stereotypes towards Aging. Snowball sampling through social media was employed, with 109 subjects completing the study.

DETAILED DESCRIPTION:
This was a quasi-experimental prospective study that used snowball sampling to recruit participants. The study was publicized through Instagram accounts of two authors with a combined following of over 100,000. Of the initial 250 participants, 109 completed the study. Inclusion criteria included:

1. Being over 18 years old.
2. Participating in both the PRE and POST questionnaires of the Negative Stereotypes towards Old Age Questionnaire (CENVE).
3. Following the Instagram posts related to the intervention for 3 days or more.

Instruments:

The evaluation instruments for this study included two online Google Forms questionnaires (See in Supplementary Material) designed for pre- and post-assessment. The pre-assessment questionnaire consisted of two sections: 16 items on sociodemographic data and 15 items from the Negative Stereotypes towards Old Age Questionnaire (CENVE) (Blanca et al., 2005). This instrument assesses individuals' stereotypes towards the older population using a Likert-type response scale ranging from 1 to 4 (1 = Strongly Disagree, 2 = Somewhat Disagree, 3 = Somewhat Agree, 4 = Strongly Agree). It provides a total score and three dimensions: Health Dimension, Social Motivation Dimension, and Character/Personality Dimension. The maximum score on this questionnaire is 60 points (indicating a high presence of negative stereotypes towards old age), and the minimum score is 15 points (indicating a low presence of such stereotypes).

Procedure:

Both at the initial and final questionnaire stages, that is, before and after the 7-day intervention period of reading the posts, was administered the questionnaire CENVE. Additionally, the post-intervention evaluation included a new question that gathered data on the frequency with which the participant had followed the intervention (0-2, 3-4, and 5-7 days).

Intervention The intervention consisted of daily positive messages about aging posted on an Instagram account (@laetapaplateada), created specifically for this study, and was conducted over the course of a week. Examples included "The ability to make decisions improves with age" and "Emotional regulation improves with age" (David, 2017). These posts were accompanied by their respective author references.

Statistical Analysis:

A paired samples t-test was conducted to compare each subject's total score on the CENVE scale before and after the intervention. To determine if certain sociodemographic variables were associated with the presence of negative stereotypes towards old age, the scores obtained in the PRE questionnaire for each study group were analyzed using descriptive statistics and hypothesis testing. This analysis was performed using Student's t-test (for variables with 2 categories) or ANOVA (for variables with more than 2 categories). The analysis of the "sex" variable was omitted due to low male participation.

Furthermore, to examine if various demographic variables were associated with pre-post differences in the presentation of negative stereotypes towards older people, a Repeated Measures ANOVA was performed for each of the sociodemographic variables collected in the questionnaires: sex, age, marital status, place of residence, cohabitants, religion, education level, occupation, frequency of contact with older people, area of contact with older people, cohabitation with older people, relationship with grandparents, significance level of that relationship, knowledge of any of their grandparents' loss of abilities (physical/mental), frequency of viewing intervention posts on Instagram, etc.

All tests were analyzed using the statistical software Jamovi 2.3.21. Data for the assessment of negative stereotypes towards old age were collected in February and March 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years old.
2. Participating in both the PRE and POST questionnaires of the Negative Stereotypes towards Old Age Questionnaire (CENVE).
3. Following the Instagram posts related to the intervention for 3 days or more.

Exclusion Criteria:

1. Being under 18 years old.
2. Participating in only one questionnaire
3. Following the Instagram posts related to the intervention for less than 3 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 109 participants over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Reduce negative stereotypes towards older people by viewing positive messages on social networks and subsequent analysis using the CENVE questionnaire | 7 days
  We use for this study two Google Forms questionnaires designed for pre- and post-assessment. There are two sections: sociodemographic data Negative Stereotypes towards Old Age Questionnaire (CENVE). The post-intervention evaluation included a new questionon the frequency with which the participant had followed the intervention. The intervention consisted of daily positive messages about aging posted on an Instagram account. The primary objective of this study was to analyze whether positive education about aging disseminated through social media could reduce negative stereotypes towards older adults. We collected data on the participants' engagement with the intervention and measure if the participants had lower scores on CENVE than before the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Zarazgoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data used to support the findings of the present study are available from the corresponding autor upon request.

REFERENCES:
- [Background] Olshansky S, Biggs S, Achenbaum W, Davison G, Fried L, Gutman G, et al. The Global Agenda Council on the Ageing Society: Policy Principles. Global Policy. 2011;2:97-105.
- [Background] World Health Organisation. Global report on ageism.
- [Background] North MS, Fiske ST. Modern Attitudes Toward Older Adults in the Aging World: A Cross-Cultural Meta-Analysis. Psychol Bull. 2015 Sep;141(5):993-1021. doi: 10.1037/a0039469. Epub 2015 Jul 20. PMID 26191955
- [Background] Levy BR, Slade MD, Chang ES, Kannoth S, Wang SY. Ageism Amplifies Cost and Prevalence of Health Conditions. Gerontologist. 2020 Jan 24;60(1):174-181. doi: 10.1093/geront/gny131. PMID 30423119
- [Background] Kornadt AE, Pauly T, Schilling OK, Kunzmann U, Katzorreck M, Lucke AJ, Hoppmann CA, Gerstorf D, Wahl HW. Momentary subjective age is associated with perceived and physiological stress in the daily lives of old and very old adults. Psychol Aging. 2022 Dec;37(8):863-875. doi: 10.1037/pag0000711. Epub 2022 Sep 22. PMID 36136787
- [Background] Nelson TD. Promoting healthy aging by confronting ageism. Am Psychol. 2016 May-Jun;71(4):276-82. doi: 10.1037/a0040221. PMID 27159434
- [Background] Hannah J. Swift. The Risks of Ageism Model: How Ageism and Negative Attitudes toward Age Can Be a Barrier to Active Aging.
- [Background] Burnes D, Sheppard C, Henderson CR Jr, Wassel M, Cope R, Barber C, Pillemer K. Interventions to Reduce Ageism Against Older Adults: A Systematic Review and Meta-Analysis. Am J Public Health. 2019 Aug;109(8):e1-e9. doi: 10.2105/AJPH.2019.305123. Epub 2019 Jun 20. PMID 31219720
- [Background] Dulcey Ruiz E, Uribe Valdivieso C. Sistema de Información Científica [Internet]. Vol. 34, Revista Latinoamericana de Psicología. Available from: http://www.redalyc.org/articulo.oa?id=80534202
- [Background] Levin JS, Chatters LM. Religion, health, and psychological well-being in older adults: findings from three national surveys. J Aging Health. 1998 Nov;10(4):504-31. doi: 10.1177/089826439801000406. PMID 10346697
- [Background] Crawford PA. Rock of Ages: Developing Healthy Perspectives of Aging in the Elementary Grades. Child Educ. 2015;91:395-401.
- [Background] Jiménez TMM. Redes sociales en prevención y promoción de la salud. Una revisión de la actualidad = Social networks in prevention and health promotion. A review of the current. REVISTA ESPAÑOLA DE COMUNICACIÓN EN SALUD. 2015 [cited 2024 Feb 1];62-9.
- [Background] Valle CG, Tate DF, Mayer DK, Allicock M, Cai J. A randomized trial of a Facebook-based physical activity intervention for young adult cancer survivors. J Cancer Surviv. 2013 Sep;7(3):355-68. doi: 10.1007/s11764-013-0279-5. Epub 2013 Mar 27. PMID 23532799
- [Background] Ridout B, Campbell A. Using Facebook to deliver a social norm intervention to reduce problem drinking at university. Drug Alcohol Rev. 2014 Nov;33(6):667-73. doi: 10.1111/dar.12141. Epub 2014 Apr 1. PMID 24689339
- [Background] Pechmann C, Delucchi K, Lakon CM, Prochaska JJ. Randomised controlled trial evaluation of Tweet2Quit: a social network quit-smoking intervention. Tob Control. 2017 Mar;26(2):188-194. doi: 10.1136/tobaccocontrol-2015-052768. Epub 2016 Feb 29. PMID 26928205
- [Background] Silfee VJ, Haughton CF, Jake-Schoffman DE, Lopez-Cepero A, May CN, Sreedhara M, Rosal MC, Lemon SC. Objective measurement of physical activity outcomes in lifestyle interventions among adults: A systematic review. Prev Med Rep. 2018 May 10;11:74-80. doi: 10.1016/j.pmedr.2018.05.003. eCollection 2018 Sep. PMID 29984142
- [Background] Alshahrani A, Siddiqui A, Khalil S, Farag S, Alshahrani N, Alsabaani A, Korairi H. WhatsApp-based intervention for promoting physical activity among female college students, Saudi Arabia: a randomized controlled trial. East Mediterr Health J. 2021 Aug 26;27(8):782-789. doi: 10.26719/emhj.21.012. PMID 34486714
- [Background] Leong CM, Lee TI, Chien YM, Kuo LN, Kuo YF, Chen HY. Social Media-Delivered Patient Education to Enhance Self-management and Attitudes of Patients with Type 2 Diabetes During the COVID-19 Pandemic: Randomized Controlled Trial. J Med Internet Res. 2022 Mar 23;24(3):e31449. doi: 10.2196/31449. PMID 35319478
- [Background] Sanchez LM, Park SY, Kohnen T, Sarnquist B, Jeon HJJ, Granner M, Morning K, MacNeil P, Deavers O, Soto V, Christiansen E. Social media intervention for promoting breastfeeding among WIC participants. Food Sci Nutr. 2023 Aug 23;11(11):6945-6954. doi: 10.1002/fsn3.3620. eCollection 2023 Nov. PMID 37970423
- [Background] Fingerman K, Trevino K. Don't Lump Seniors Together on Coronavirus. Older People Aren't All the Same. USA Today. 2020 Apr 7.
- [Background] Wahl H-W, Gerstorf D. A conceptual framework for studying Context Dynamics in Aging (CODA). Dev Rev. 2018;50(Part B):155-176.
- [Background] Sanchez Palacios C, Trianes Torres MV, Blanca Mena MJ. [Aging negative stereotypes and their relationship with sociodemographic variables over 65 elderly]. Rev Esp Geriatr Gerontol. 2009 May-Jun;44(3):124-9. doi: 10.1016/j.regg.2008.12.008. Epub 2009 May 14. Spanish. PMID 19446376
- [Background] Menendez Alvarez-Dardet S, Cuevas-Toro AM, Perez-Padilla J, Lorence Lara B. [Assessment of negative stereotypes about old age in young people and adults]. Rev Esp Geriatr Gerontol. 2016 Nov-Dec;51(6):323-328. doi: 10.1016/j.regg.2015.12.003. Epub 2016 Jan 28. Spanish. PMID 26826942
- [Background] Antonio Hidalgo Sacristán. Estereotipos edadistas en una muestra de adultos jóvenes.
- [Background] Colás P, Villaciervos P. La interiorización de los estereotipos de género en jóvenes y adolescentes. Revista de Investigación Educativa. 2007;25(1).
- [Background] Kim HH, Jung JH. Ageism, Religiosity, and Wellbeing Among Older Adults: Evidence From the European Social Survey (ESS4). Res Aging. 2021 May;43(5-6):214-226. doi: 10.1177/0164027520953632. Epub 2020 Sep 2. PMID 32873186
- [Background] Stevens-Long J, Michaud G. THEORY IN ADULT DEVELOPMENT: The New Paradigm and the Problem of Direction.
- [Background] Officer A, de la Fuente-Nunez V. A global campaign to combat ageism. Bull World Health Organ. 2018 Apr 1;96(4):295-296. doi: 10.2471/BLT.17.202424. Epub 2018 Mar 9. No abstract available. PMID 29695887
- [Background] Coq D, Rosario H, Chaves A. Metodología de Encuestas A EMPRESARIOS ANDALUCES. 2002 [cited 2024 Feb 1];4:211-25.
- [Derived] Fuente-Hernandez L, de la Fuente-Ruiz E, Gracia-Garcia P, Serrano-Garcia I, Alvarez-Mon MA, Molina-Ruiz RM. Using social media-based positive education to challenge negative stereotypes of aging: a quasi-experimental approach. BMC Public Health. 2025 Feb 10;25(1):533. doi: 10.1186/s12889-025-21327-0. PMID 39930436

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT06574243/Prot_SAP_ICF_000.pdf